CLINICAL TRIAL: NCT02406911
Title: Relationship of Dose of Ticagrelor and Anti-inflammatory Effect in Patients With End Stage Renal Disease on Hemodialysis: PIANO-6 Randomized Crossover Study
Brief Title: Ticagrelor and Anti-inflammatory Effects
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Weon Kim, Professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PIANO6
Record Dates: First submitted 2015-03-14; First posted 2015-04-02 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Kidney Disease
Keywords: platelet; ticagrelor; clopidogrel; end stage renal disease; hemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor 90 mg (Experimental): After randomization, an initial loading dose of ticagrelor (180 mg) was given and low dose ticagrelor (ticagrelor 90 mg once a day) was treated for 14 days.
  Interventions: Drug: Ticagrelor
- Ticagrelor 180 mg (Active Comparator): After randomization, an initial loading dose of ticagrelor (180 mg) was given and usual dose ticagrelor (ticagrelor 90 mg twice a day) was treated for 14 days.
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor — After randomization, each group will be treated as assigned dose of ticagrelor (ticagrelor 90mg once a day or 90mg twice a day) for 14 days. After 1 week wash-out period, cross-over study will be performed
  Other Names: Ticagrelor (Brilinta)

SUMMARY:
Antiplatelet treatment in patients with end stage renal disease (ESRD) on hemodialysis (HD) is still challenging because of bleeding and thrombotic complications. The investigators hypothesized ticagrelor once daily dose would achieve tolerable antiplatelet effects compared with ticagrelor twice a day dose in ESRD patients on HD.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a strong risk factor for cardiovascular morbidity and mortality, and confers an increasing risk of stent thrombosis even when dual antiplatelet therapy (clopidogrel and aspirin) is administered. Patients with severe CKD or end stage renal disease (ESRD) on hemodialysis (HD) exhibited higher platelet reactivity to clopidogrel than did those with normal renal function. The investigators recently reported platelet inhibition by ticagrelor was faster and markedly greater than by clopidogrel with onset dosing regimen in patients with ESRD on HD. However, few studies have been conducted whether platelet reactivity during ticagrelor treatment is associated with endothelial function, platelet activation markers and inflammation status in ESRD patients on HD. Additionally, the dose dependent effects of ticagrelor have been rarely evaluated.

ELIGIBILITY:
Inclusion Criteria:

* ESRD patients undergoing regular (≥ 6 months) maintenance HD
* ongoing (≥ 2 months) treatment with clopidogrel
* P2Y12 reaction units (PRUs) were more than 235

Exclusion Criteria:

* known allergies to aspirin, clopidogrel, or ticagrelor
* concomitant use of other antithrombotic drugs (oral anticoagulants, dipyridamole)
* thrombocytopenia (platelet count <100,000/mm3)
* hematocrit <25%
* uncontrolled hyperglycemia (hemoglobin A1c >10%)
* liver disease (bilirubin level >2 mg/dl)
* symptomatic severe pulmonary disease
* active bleeding or bleeding diathesis
* gastrointestinal bleeding within the last 6 months
* hemodynamic instability
* acute coronary or cerebrovascular event within the last 3 months
* pregnancy
* any malignancy
* concomitant use of a cytochrome P450 inhibitor or nonsteroidal anti-inflammatory drug
* recent treatment (<30 days) with a glycoprotein IIb/IIIa antagonist

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-06 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
The difference of antiplatelet effects assessed by VerifyNow assay | 14 days after study drug treatment
  The difference of PRU values achieved following antiplatelet therapy

SECONDARY OUTCOMES:
The difference of antiplatelet effects assessed by light aggregometry assay | 14 days after study drug treatment
  The difference of IPA values achieved following antiplatelet therapy
The difference of endothelial function assessed by forearm flow-mediated vasodilation (FMD) and peripheral arterial tonometry (PAT) | 14 days after study drug treatment
  The difference of endothelial functions achieved following antiplatelet therapy
The difference of anti-inflammatory biomarkers | 14 days after study drug treatment
  The difference of hsCRP, CD40, P-selectin, and IL-6

OTHER OUTCOMES:
Adverse events | 6 weeks
  Adverse events such as bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Weon kim, MD, PhD, Principal Investigator — Kyung Hee University Hospital
Locations (1):
- Kyung Hee University Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730